CLINICAL TRIAL: NCT00941668
Title: Evaluate Inflammation Caused by Gingivitis in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-1005-INF-UNC-FP
Record Dates: First submitted 2008-09-26; First posted 2009-07-17 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Toothpaste (Active Comparator): Triclosan/Copolymer/fluoride toothpaste
  Interventions: Drug: Triclosan/Copolymer/fluoride toothpaste
- Fluoride toothpaste (Placebo Comparator): sodium monofluorophosphate toothpaste
  Interventions: Drug: sodium monofluorophosphate toothpaste

INTERVENTIONS:
Drug: Triclosan/Copolymer/fluoride toothpaste — Twice daily usage
  Other Names: Total toothpaste
  Arms: Total Toothpaste
Drug: sodium monofluorophosphate toothpaste — Twice daily usage
  Other Names: Colgate cavity protection toothpaste
  Arms: Fluoride toothpaste

SUMMARY:
The purpose of this study is to compare the anti-inflammatory efficacy of a dentifrice

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adult males or females 18 to 60 years old
* Subjects must be able and willing to follow study procedures and instructions
* Subjects must have generalized, moderate plaque-associated gingivitis as determined by the Investigator or designee during the screening examination
* Subjects must present with at least 20 teeth in the functional dentition, excluding third molars
* Each subject must have at least four teeth with probing depths of 4-5 millimeters and at least 30% of sites bleeding to gentle probing

Exclusion Criteria:

* Subjects who have chronically used (two weeks or more) Total (Triclosan/Copolymer) dentifrice within 6 months prior to enrollment
* Subjects with gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque and calculus, or soft or hard tissue tumor of the oral cavity
* Subjects with periodontitis as indicated by periodontal pocketing 6 millimeters at screening
* Subjects with a history of early onset periodontitis or acute necrotizing ulcerative gingivitis
* Subjects with concomitant endodontic or periodontal therapy other than prophylaxis within 6 months prior to enrollment
* Subjects with orthodontic appliances or removable partial dentures
* Subjects chronically treated (two weeks or more) with any medication known to affect inflammation or periodontal status or (aspirin, nonsteroidal anti-inflammatory drugs, steroids, statins, phenytoin, calcium antagonists, cyclosporin and coumadin) within one month of the screening examination. All other medications for chronic medical conditions should be initiated at least three months prior to enrollment
* Subjects who currently smoke or who report using tobacco products within one year of screening.
* Subjects who have been treated with antibiotics for medical or dental reasons within 3 months prior to enrollment
* Subjects having clinically significant or unstable organic disease; subjects having compromised healing potential such as those with diabetes mellitus or connective tissue disorders; subjects having heart murmurs, histories of rheumatic fever, valvular disease or prosthetic joint replacement necessitating antibiotic prophylaxis
* Female subjects who report being pregnant
* Subjects who use hormonal contraceptives must have started the method 30 days prior to the screening examination.
* Subjects with active infectious diseases such as hepatitis, human immunodeficiency virus or Tuberculosis
* Subjects diagnosed with human immunodeficiency virus (HIV) or subjects that are immunocompromised as determined by the Investigator
* Medical condition which precludes not eating/drinking for approximately 8 hours.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Paquette, DMD, Principal Investigator
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited by the PI at the clinical site
Groups:
- Total Toothpaste (Active): triclosan/copolymer/fluoride toothpaste
- Colgate Great Regular Flavor (Placebo): sodium monofluorophosphate toothpaste
Period: Overall Study
Arm/Group | Total Toothpaste (Active) | Colgate Great Regular Flavor (Placebo)
Started | 24 | 25
Completed | 0 | 0
Not Completed | 24 | 25

BASELINE CHARACTERISTICS:
Groups:
- Colgate Cavity Protection (Placebo): sodium monofluorophosphate toothpaste
- Total: Total of all reporting groups
Arm/Group | Total Toothpaste (Active) | Colgate Cavity Protection (Placebo) | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (12.5) | 34 (12.1) | 36.25 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Level of Gingival Crevicular Fluid Interleukin - 1 (GCF IL-1) at 2 Hours
Description: Levels of Gingival crevicular fluid Interleukin - 1 (GCF IL-1)(weight in micrograms)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | Total Toothpaste (Active) | Colgate Cavity Protection (Placebo)
Number analyzed (Participants) | 24 | 25
Micrograms | 492.2 (545.5) | 326.3 (307.7)
Statistical Analysis 1: Comparison: Total Toothpaste (Active) vs Colgate Cavity Protection (Placebo); The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Primary Outcome: Level of Gingival Crevicular Fluid Interleukin - 6(GCF IL-6) at 2 Hours
Description: Levels of Gingival crevicular fluid Interleukin - 6 (GCF IL-6) (weight in micrograms)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | Total Toothpaste (Active) | Colgate Cavity Protection (Placebo)
Number analyzed (Participants) | 24 | 25
Micrograms | 12.8 (23.3) | 21.3 (46.4)
Statistical Analysis 1: Comparison: Total Toothpaste (Active) vs Colgate Cavity Protection (Placebo); The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | Total Toothpaste (Active) | Colgate Cavity Protection (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 1/24 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Toothpaste (Active) (N=24) | Colgate Cavity Protection (Placebo) (N=25)
Tooth Sensitivity to Cold (General disorders) | 1 (1) | 2 (2) — Subjects reported tooth sensitivity to cold
Oral irritation (General disorders) | 1 (1) | 1 (1) — subject reported oral irritation after using the study product
Cold and/or flu like symptoms (General disorders) | 1 (1) | 2 (2) — 2 subjects reported cold like symptoms halfway through the study and 1 subject reported flu like symptoms (Fever,chills and sore throat) at end of study.
pulled muscle (General disorders) | 1 (1) | 1 (1) — 1 subject reported a pulled muscle in their back at the end of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days